CLINICAL TRIAL: NCT04583631
Title: Relationship Between Apoptosis and er Stress in Chronic Adenoiditis and Adenoid Hypertrophy
Brief Title: Relationship of Endoplasmic Reticulum Stress and Adenoid Diseases
Status: Completed | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Merih Onal, Assistant Professor, Selcuk University
Other Study IDs: 2018-18
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Adenoiditis Acute Infective
Keywords: Adenoidectomy; ; Endoplasmic Reticulum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Adenoid tissues were gathered in groups in accordance with their size and analyzed in regards to ER stress and apoptosis markers by Real-Time PCR and Western Blotting method.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic adenoiditis: Patients with hypertrophy and those out of hypertrophy were determined and those who had purulant rhinorrhea signs and rate of adenoids-choana below 50% were categorized that chronic adenoiditis.
  Interventions: Procedure: Adenoidectomy surgery
- Adenoid hypertrophy: Patients who have snoring and those whose adenoid choana rate is greater than 50% were categorized that adenoid hypertrophy group.
  Interventions: Procedure: Adenoidectomy surgery

INTERVENTIONS:
Procedure: Adenoidectomy surgery — All patients underwent adenoidectomy under general anesthesia by routine curettage method and adenoid tissues were put in formaldehyde and sent to the genetics department for the exploration of ER stress and apoptosis markers.

SUMMARY:
Adenoid tissue is a significant organ for the performing of immune systems in children. The Endoplasmic Reticulum (ER), is an organelle needed for the care of a stable function of cells. The purpose of the study was to explore the correlation among ER stress and adenoid tissue disorders and to explain the structure of diseases related to the immune system.

ELIGIBILITY:
Inclusion Criteria:

- Patients with the clinical diagnosis of chronic adenoiditis and adenoid hypertrophy.

Exclusion Criteria:

* Systemic diseases
* Other otolaryngological

Ages: 3 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study was performed on 54 patients (28 male, 26 female) between the ages of 3 and 9 (mean 5) with the clinical diagnosis of chronic adenoiditis and adenoid hypertrophy and who underwent adenoidectomy due to either chronic adenoiditis or adenoid hypertrophy.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Correlation of ER stress and apoptosis with chronic adenoiditis and adenoid hypertrophy | 2018-2019 (1 year)
  Our primary outcome was to evaluate providing that ER stress and apoptosis reaction performing in chronic adenoiditis and adenoid hypertropy, which is related with the immune system of children.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Selcuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
We will share study protocol after our article has been accepted for publication in a journal.

REFERENCES:
- [Background] Casselbrant ML. What is wrong in chronic adenoiditis/tonsillitis anatomical considerations. Int J Pediatr Otorhinolaryngol. 1999 Oct 5;49 Suppl 1:S133-5. doi: 10.1016/s0165-5876(99)00147-0. PMID 10577791
- [Background] Li R, Wang Y, Chen P, Meng J, Zhang H. Inhibiting endoplasmic reticulum stress by activation of G-protein-coupled estrogen receptor to protect retinal astrocytes under hyperoxia. J Biochem Mol Toxicol. 2021 Feb;35(2):e22641. doi: 10.1002/jbt.22641. Epub 2020 Sep 29. PMID 32996202